CLINICAL TRIAL: NCT02734355
Title: Upstream-therapy by Telmisartan and Amlodipine Combination for Improvement of Left Atrial Mechanical Function After Pulmonary Vein Antrum Isolation
Brief Title: Left Atrial Mechanical Function Improvement After Atrial Fibrillation Catheter Ablation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Research Institute for Complex Problems of Cardiovascular Diseases, Russia (Other)
Responsible Party: Principal Investigator, Sergey Mamchur, Head of Department of Cardiovascular Disorders Diagnosis, Research Institute for Complex Problems of Cardiovascular Diseases, Russia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0546-2015-0013
Record Dates: First submitted 2016-03-30; First posted 2016-04-12 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; left atrium; mechanical function; contractility
MeSH Terms: conditions — Atrial Fibrillation | interventions — Telmisartan; Amlodipine; telmisartan amlodipine combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapy (Active Comparator): Telmisartan 80 mg and amlodipine 5 mg tablet by mouth every 24 hours for 7 days
  Interventions: Drug: Telmisartan 80 mg and amlodipine 5 mg
- Placebo (Placebo Comparator): Placebo (for telmisartan 80 mg and amlodipine 5 mg) tablet by mouth every 24 hours for 7 days
  Interventions: Drug: Placebo (for telmisartan and amlodipine)

INTERVENTIONS:
Drug: Telmisartan 80 mg and amlodipine 5 mg
  Other Names: Twynsta
  Arms: Therapy
Drug: Placebo (for telmisartan and amlodipine) — Sugar pill manufactured to mimic telmisartan 80 mg and amlodipine 5 mg tablet
  Arms: Placebo

SUMMARY:
The objective of the study was to estimate the efficacy of telmisartan and amlodipine combination on the restoration of left atrial mechanical function after atrial fibrillation catheter ablation.

DETAILED DESCRIPTION:
64 candidates to atrial fibrillation ablation were included in the study. Patients were randomly assigned to telmisartan/amlodipine combination in dose 80/5 mg (group I, n=34) or placebo (group II, n=30) taking daily for up to one week. Echocardiography was performed before the procedure, immediately after it, and after a week of therapy. The six-minute walk test and SF-36 questionnaire results were evaluated a day before the procedure and after a week of the therapy. The left ventricular end-diastolic pressure was invasively measured after transseptal puncture and before left atrial sheath removal.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic (III-IV class by European Heart Rhythm Association scale) paroxysmal atrial fibrillation;
* Ineffective therapy by at least one of the class I or III antiarrhythmic drugs;
* Left atrial diameter 5 cm or less;
* Estimated catheter radiofrequency pulmonary vein antrum isolation;
* Signed informed consent.

Exclusion Criteria:

* Intolerance/allergy or contraindications to telmisartan, amlodipine, warfarin or enoxaparin;
* Left atrial thrombosis;
* Age greater than 75 years;
* Severe (e.g. decompensation of vital functions) or acute (e.g. pneumonia) somatic conditions;
* Malignant growth in the hematogenic dissemination stage.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yevgeny V Grigoriev, M.D., Ph.D., Study Chair — Research Institute for Complex Problems of Cardiovascular Diseases

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mamchur S, Mamchur I, Khomenko E, Kokov A, Bokhan N, Sherbinina D. Mechanical function of left atrium and pulmonary vein sleeves before and after their antrum isolation. Medicina (Kaunas). 2014;50(6):353-9. doi: 10.1016/j.medici.2014.11.008. Epub 2014 Nov 28. PMID 25541269

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Therapy | Placebo
Started | 34 | 30
Completed | 34 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Therapy: Telmisartan 80 mg and amlodipine 5 mg tablet by mouth every 24 hours for 7 days
  Telmisartan 80 mg and amlodipine 5 mg
- Total: Total of all reporting groups
Arm/Group | Therapy | Placebo | Total
Number analyzed (Participants) | 34 | 30 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (5.7) | 54.1 (6.2) | 53.1 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 22 | 19 | 41
Region of Enrollment [Count of Participants; unit: Participants]
  Russian Federation | 34 | 30 | 64

OUTCOME MEASURES:

1. Primary Outcome: Passive Emptying of Left Atrium
Description: Velocity time integral of transmitral flow during left ventricle early filling phase (VTI E, cm).
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Therapy | Placebo
Number analyzed (Participants) | 34 | 30
cm | 14.7 (4.4) | 20.9 (5.2)

2. Primary Outcome: Active Emptying of Left Atrium
Description: Velocity time integral of transmitral flow during atrial contraction (VTI A, cm).
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Therapy | Placebo
Number analyzed (Participants) | 34 | 30
cm | 7.4 (2.6) | 5.4 (1.3)

3. Primary Outcome: Left Atrial Reservoir Function
Description: Velocity time integral of transmitral flow (VTITMF, cm) during the whole diastole.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Therapy | Placebo
Number analyzed (Participants) | 34 | 30
cm | 19.1 (3.5) | 13.3 (3.2)

4. Primary Outcome: Diastolic Function
Description: E/A ratio of transmitral flow
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Therapy | Placebo
Number analyzed (Participants) | 34 | 30
ratio | 1.62 (0.35) | 2.64 (0.63)

5. Primary Outcome: Isovolumic Relaxation
Description: Left ventricular isovolumic relaxation time (IVRT, ms).
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Therapy | Placebo
Number analyzed (Participants) | 34 | 30
ms | 117 (19) | 98 (10)

6. Primary Outcome: Pulmonary Vein Flow Emptying
Description: S/D ratio of right superior pulmonary vein flow
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Therapy | Placebo
Number analyzed (Participants) | 34 | 30
ratio | 1.3 (0.39) | 1.46 (0.37)

7. Primary Outcome: Retrograde Flow in Pulmonary Veins
Description: Velocity time integral of right superior pulmonary vein flow during left atrial systole (VTI Ar, cm)
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Therapy | Placebo
Number analyzed (Participants) | 34 | 30
cm | 4.1 (1.4) | 1.5 (0.5)

8. Primary Outcome: Left Atrial Contractility
Description: Left atrial active emptying fraction (LAAEF, %)
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: percentage of LA maximum volume
Arm/Group | Therapy | Placebo
Number analyzed (Participants) | 34 | 30
percentage of LA maximum volume | 40 (6.7) | 31.6 (6.7)

9. Primary Outcome: Left Atrial Dimensions
Description: Left atrial antero-posterior diameter (LAD, cm)
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Therapy | Placebo
Number analyzed (Participants) | 34 | 30
cm | 3.9 (0.3) | 4.1 (0.6)

10. Primary Outcome: Left Atrial Pressure Load
Description: Mean left atrial pressure (MLAP, mm Hg).
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Therapy | Placebo
Number analyzed (Participants) | 34 | 30
mm Hg | 9 (3.1) | 13.8 (2.9)

11. Primary Outcome: Pulmonary Circulation Pressure Load
Description: Right ventricular systolic pressure (RVSP, mm Hg).
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Therapy | Placebo
Number analyzed (Participants) | 34 | 30
mm Hg | 16.7 (9.6) | 31.6 (14.4)

12. Secondary Outcome: Quality of Life
Description: The average of eight scores of 36-Item Short Form Health Survey (SF-36). In every case all of eight scores (which ranges from 0 to 100) was summarized, then the sum was divided by 8. Thus the outcome also ranges from 0 (worse outcome) to 100 (better outcome).
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapy | Placebo
Number analyzed (Participants) | 34 | 30
units on a scale | 92 (4) | 85 (5)

13. Secondary Outcome: Exercise Tolerance
Description: six-minute walk distance in meters
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Therapy | Placebo
Number analyzed (Participants) | 34 | 30
m | 403 (27) | 345 (25)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Therapy | Placebo
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/30
Other Adverse Events (participants affected / at risk) | 3/34 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapy (N=34) | Placebo (N=30)
Drug-induced hypotension (Cardiac disorders) | 2 (2) | 1 (1)
Swelling of lower leg (Blood and lymphatic system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes